CLINICAL TRIAL: NCT04026347
Title: An Evaluation of the Vesair® Bladder Control System for the Treatment of Stress Urinary Incontinence in Post-Menopausal Women
Brief Title: Vesair Clinical Trial
Acronym: VAPOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Missed endpoint
Sponsor: Solace Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD1010
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Stress Urinary Incontinence
Keywords: SUI; Women; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject and assessor blinded to randomization result
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Vesair (Experimental): Subjects are treated with Vesair Balloon at enrollment (day 0)
  Interventions: Device: Vesair Balloon
- Sham (Sham Comparator): Subjects are treated with sham at enrollment (day 0) and treated with balloon (if desired) after six month visit.
  Interventions: Device: Vesair Balloon; Other: Sham balloon placement

INTERVENTIONS:
Device: Vesair Balloon — Indwelling, intravesical balloon
Other: Sham balloon placement — Sham balloon placement procedure
  Arms: Sham

SUMMARY:
Single-blind, multicenter, randomized clinical trial of the Vesair Balloon in the treatment of Stress Urinary Incontinence in post-menopausal women

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with SUI for at least 12 months
* Average of at least one leak per day
* Failed non-invasive treatment
* Willing to undergo cystoscopy and a minimum of 5 visits over one year

Exclusion Criteria:

* BMI > 40.0
* Last menstrual period within 12 months of enrollment
* On birth control and/or oral hormone replacement therapy
* Urge-predominant mixed incontinence
* SUI due to intrinsic sphincter deficiency
* Prior treatment with the Vesair Balloon
* Prior medical, surgical or non-surgical treatment for SUI within 6 months of enrollment
* Recurrent or recent (within the past 5 years) kidney stones
* Recurrent or recent (within the past 3 months) Urinary Tract Infection
* Stage 3 or higher cystocele (POP-Q)
* Interstitial or follicular cystitis / painful bladder syndrome
* Local genital infection
* Artificial sphincter
* Anatomic abnormalities which would interfere with device placement.
* Visible blood in the urine
* Uncontrolled bladder contractions / discomfort with bladder filling up to 300cc
* History of cancer of the urinary tract
* History of any cancer within the past two years (excluding non-melanoma skin cancers)
* History of any cancer not (yet) treated with curable intent (excluding non-melanoma skin cancers)
* Immunologically suppressed or immunocompromised
* Undergoing pelvic radiation, pelvic fibrosis from previous pelvic radiation
* Non ambulatory / unable to do simple pad weight testing exercises
* On anticoagulation therapy with the exception of aspirin
* History of mental illness requiring inpatient treatment
* Neurological disease such as Parkinson's or multiple sclerosis
* Uncontrolled diabetes (A1C > 9%)
* Recent alcohol or drug abuse requiring treatment in the past year
* Autoimmune or connective tissue disorders such as Marfan syndrome, Ehlers-Danlos or Myasthenia Gravis
* Allergy to polyurethane or perfluorocarbons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint | 6 months
  Pad weight + I-QOL

SECONDARY OUTCOMES:
Pad Weight | 6 months
  Reduction in pad weight
I-QOL | 6 months
  Improvement in I-QOL score (0-100 point scale, 100 being the best outcome)
Episode Frequency | 6 months
  Reduction in episode frequency as reported on a 7 day diary
Patient Global Impression of Improvement (PGI-I) | 6 months
  Significant Improvement per PGI-I (response of very much better or much better on 7 point scale)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Valley Urogynecology Associates, Phoenix, Arizona
  - Scripps Clinic, San Diego, California
  - Tri Valley Urology, Temecula, California
  - Dr. Sherry Thomas, Westlake Village, California
  - Women's Health Specialty Care, Farmington, Connecticut
  - Florida Urology Partners, Tampa, Florida
  - Meridian Clinical Research / Urological Associates of Savannah, Savannah, Georgia
  - WomanCare, Arlington Heights, Illinois
  - CMB Research / Basinski and Juran MDs, Newburgh, Indiana
  - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology, Hanover, Maryland
  - Chesapeake Urology, Owings Mills, Maryland
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Mercy Health, Ada, Michigan
  - Freedman Urology, Las Vegas, Nevada
  - ProHEALTH Garden City Urology, Garden City, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - MetroHealth, Cleveland, Ohio
  - Penn Medicine, Philadelphia, Pennsylvania
  - Women and Infants dept of Urogynecology, Providence, Rhode Island
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - Washington Urology, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCammon K, Jacoby K, Kalota S, Snyder J, Cline K, Robertson K, Rardin C, Kahan R, Green L, Zuckerman J, Rovner E. Three-month primary efficacy data for the SUCCESS Trial; a phase III, multi-center, prospective, randomized, controlled study treating female stress urinary incontinence with the vesair intravesical balloon. Neurourol Urodyn. 2018 Jan;37(1):440-448. doi: 10.1002/nau.23324. Epub 2017 Nov 2. PMID 29095516
- See also: Company Website — http://www.solacetx.com